CLINICAL TRIAL: NCT05737420
Title: Video-call Assisted Assessment of Acute Stroke in Addition to Stroke Severity Scales in a Prehospital Setting: A Cluster Randomised Pilot Trial
Brief Title: Video-call Assisted Assessment of Acute Stroke in Addition to Stroke Severity Scales in a Prehospital Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHS-Neuro-1-2023
Record Dates: First submitted 2023-02-06; First posted 2023-02-21 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Stroke; Nervous System Diseases; Vascular Diseases
MeSH Terms: conditions — Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Stroke; Nervous System Diseases; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional video call (Experimental): All patients suspected of stroke in a prehospital setting are examined according to a prehospital stroke score. The emergency services personnel then contact the on-call neurologist and a live video stream is initiated. The on-call neurologist then examines the patient via the video-call.
  Interventions: Diagnostic Test: Video call
- Control with standard care (No Intervention): All patients suspected of stroke in a prehospital setting are examined according to a prehospital stroke score. The emergency services personnel then contact the on-call neurologist by telephone. .

INTERVENTIONS:
Diagnostic Test: Video call — The on-call neurologist can see and communicate with the patient via live stream video-call.
  Arms: Interventional video call

SUMMARY:
This study aims to investigate whether a live stream video between the on-call neurologist and the emergency medical services is feasible.

DETAILED DESCRIPTION:
Multiple stroke severity scales have been coined in order to examine patients suspected of stroke in a prehospital setting in order to identify and transfer patients eligible for thrombectomy directly to a comprehensive stroke centre (CSC). However, performance and feasibility vary greatly in different validation studies suggesting that those outcomes are greatly dependent on other factors i.e. acceptance amongst stakeholders, implementation process, patient segment etc. Some recent studies have shown promising results using telemedicine i.e. video solutions between emergency medical services (EMS) personnel and on-call neurologist in examining patients suspected of stroke in the prehospital phase. The investigators will perform this trial to examine whether a cluster randomised trial with video call assisted assessment of patients suspected of stroke in a prehospital setting is an appropriate trial design and feasible with regard to recruitment and retention, acceptability among stakeholders (EMS and neurologists) as well as patients and lastly with regard to stakeholders' adherence to protocol.

ELIGIBILITY:
Inclusion Criteria:

* Suspected stroke within 24 hours from onset (confirmed with Pre-hospital stroke score 1 ≥1)
* Catchment area of Hospital Sønderjylland
* Deferred informed consent obtained from patient or patient surrogate

Exclusion Criteria:

* In-hospital stroke or private transport to hospital
* Unconsciousness defined as Glascow Coma Score (GCS) ≤ 8 (as they cannot be rated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | Through study completion, approximately 2 months
  Rate of patients included in the trial amongst all patients screened
Exclusion rate | Through study completion, approximately 2 months
  rate of patients excluded from participation amongst all patients screened
Attrition rate | Through study completion, approximately 5 months
  rate of patients and data lost
Adherence to protocol by the Emergency Medical Services | Baseline (Prehospital examination of patient conducted by Emergency Medical Services)
  Evaluation of missing data in the clinical examination prehospital in Pre-hospital patient journal
Adherence to protocol by the neurologist prehospital | Baseline (Prehospital examination of patient conducted on video by neurologists)
  Evaluation of missing data in the clinical examination conducted with video
Adherence to protocol by the neurologist intrahospital | At admission
  Evaluation of missing data in the National Institute of Health Stroke Scale conducted intrahospital by neurologist
Stakeholder Feedback Survey | immediately after the intervention
  Mixed open-ended and closed (Likert type response) questions to assess trial and intervention acceptability
Patient Feedback Survey | Between the day after admission and 5 days after admission
  Semistructured interview with open-ended and closed (Likert type response) questions to assess intervention acceptability

SECONDARY OUTCOMES:
Acute ischemic stroke with Large Vessel Occlusion on neuroimaging | At admission
  Acute ischemic stroke with Large Vessel Occlusion (LVO) on neuroimaging (computer tomography (CT), CT angiography, magnetic resonance imaging (MRi), MR angiography or catheter-based angiography). LVO is defined as an occlusion or sub-occlusion of the intracranial internal carotid artery, middle cerebral artery M1 or M2, basilar artery. Sign of a dense cerebral artery on CT is also considered LVO positive.
Other large vessel Acute ischemic stroke | at admission
  Neuroimaging (computer tomography (CT), CT angiography, magnetic resonance imaging (MRi), MR angiography or catheter-based angiography) with AIS with occlusion or sub-occlusion of either anterior cerebral artery A1 or A2, posterior cortical artery P1 or intracranial vertebral artery
Other Acute ischemic stroke | at admission
  Neuroimaging (computer tomography (CT), CT angiography, magnetic resonance imaging (MRi), MR angiography or catheter-based angiography) with Acute ischemic stroke
Haemorrhagic stroke | at admission
  Neuroimaging (computer tomography (CT), CT angiography, magnetic resonance imaging (MRi), MR angiography or catheter-based angiography) with intra cranial haemorrhage (ICH)
Duration of examination on video-call | up to 60 minutes (prior to admission, prehospital phase)
  Duration of examination on video-call measured in minutes
Mimic mistaken for stroke | Through study completion, approximately 2 months
  Mimic mistaken for stroke evaluated as discrepancy between stroke as tentative diagnoses at primary contact from EMS and final diagnosis at discharge
Prehospital time on scene | up to 60 minutes (at prehospital contact)
  Time on scene from arrival of Emergency Medical Services to departure of Emergency Medical Services measured in minutes
90 days modified Rankin Scale | 90 days post admission date
  Modified Rankin Scale score in stroke patients as evaluated through a structured telephone-based interview performed by a central assessor who is blinded to group assignment

CONTACTS AND LOCATIONS:
Overall Officials: Christian Backer Mogensen, Study Director — Hospital of Southern Denmark - Aabenraa
Locations (1):
- Sygehus Soenderjylland, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen TTM, van den Wijngaard IR, Bosch J, van Belle E, van Zwet EW, Dofferhoff-Vermeulen T, Duijndam D, Koster GT, de Schryver ELLM, Kloos LMH, de Laat KF, Aerden LAM, Zylicz SA, Wermer MJH, Kruyt ND. Comparison of Prehospital Scales for Predicting Large Anterior Vessel Occlusion in the Ambulance Setting. JAMA Neurol. 2021 Feb 1;78(2):157-164. doi: 10.1001/jamaneurol.2020.4418. PMID 33252631
- [Background] Mazya MV, Berglund A, Ahmed N, von Euler M, Holmin S, Laska AC, Mathe JM, Sjostrand C, Eriksson EE. Implementation of a Prehospital Stroke Triage System Using Symptom Severity and Teleconsultation in the Stockholm Stroke Triage Study. JAMA Neurol. 2020 Jun 1;77(6):691-699. doi: 10.1001/jamaneurol.2020.0319. PMID 32250423